CLINICAL TRIAL: NCT04699305
Title: An Observational Clinical Registry to Collect Safety and Efficacy Data on Wound Care in Medical Centers
Brief Title: Safety and Efficacy of ActiGraft Treatment in Wound Care in Medical Centers
Status: Recruiting | Type: Observational
Sponsor: RedDress Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RD005
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cutaneous Wounds
Keywords: DFU, PU, Surgical, Vascular, Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- ActiGraft: Whole blood clot (WBC) gel
  Interventions: Device: ActiGraft

INTERVENTIONS:
Device: ActiGraft — Whole blood clot (WBC) gel

SUMMARY:
Multicenter observational study to explore the efficacy of ActiGraft in the treatment of exuding cutaneous wounds in real-life usage.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Subject has an exuding cutaneous wound
* Subject agrees to the use of his health data, including photos of his wound in analysis and publications
* Subject/LAR must be able to read and understand English and/or Spanish

Exclusion Criteria:

* Subject/LAR is unable to read and understand English or Spanish.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with all types of exuding cutaneous wound
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage area reduction (PAR) at 4 weeks | 4 weeks
  Change from baseline at 4 weeks of wounds treated with ACTIGRAFT compared to other treatments (no ACTIGRAFT).
Nature, frequency, and severity of adverse events in the intent to treat population | 1 year
  Nature, frequency, and severity (by CTCAE5) of adverse events

SECONDARY OUTCOMES:
Percentage area reduction at 8 and 12 weeks | 12 weeks
  Change from baseline at 8 and 12 weeks of wounds treated with ACTIGRAFT compared to other treatments (no ACTIGRAFT).

OTHER OUTCOMES:
Reduction in pain at 4 weeks | 4 weeks
  Pain reduction at 4 weeks for wounds treated with ACTIGRAFT compared to other treatments (no ACTIGRAFT) for patients reporting any level of wound related pain (>1 on a VAS scale of 0-10 points) at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Sirota, Study Director — RedDress Ltd.
Locations (1):
- Wound Care Experts, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
The results will be part of several scientific publications
Supporting Information: Study Protocol
Time Frame: Upon publication

REFERENCES:
- [Derived] Williams M, Davidson D, Wahab N, Hawkins J, Wachuku CD, Snyder R. Innovative treatment utilizing an autologous blood clot for diabetic foot ulcers. Wounds. 2022 Jul;34(7):195-200. doi: 10.25270/wnds/21089. PMID 35881826